CLINICAL TRIAL: NCT04598815
Title: A Phase II, Randomized, Superiority, Adaptive, Open-label, Single-center, Clinical Trial to Evaluate the Efficacy of Sirolimus (Rapamycin) in Patients With Graves' Disease and Moderate-to-severe and Active Graves' Orbitopathy (GO)
Brief Title: Sirolimus for Graves' Orbitopathy (GO)
Acronym: SIRGO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Associate Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIRGO
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus (Experimental): Sirolimus for 12 weeks
  Interventions: Drug: Sirolimus
- Methylprendnisolone (Experimental): Methylprednisolone for 12 weeks
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Group Sirolimus: Patients will receive a first dose of Sirolimus of one 2 mg tablet on the first day, given approximately at 10 am, followed by 0.5 mg tablet per day for 12 weeks.
  Group Methylprednisolone: Methylprednisolone pulse therapy will be administered for 12 weeks as follows: 500 mg iv once weekly for 6 weeks, then 250 mg iv once weekly for a further 6 weeks, for a cumulative dose 4.5 g.
  Other Names: Rapamycin

SUMMARY:
Graves' Orbitopathy (GO) is a disabling and disfiguring condition associated with Graves' Disease, due to autoimmunity against antigens expressed by the thyroid and orbital tissues, and resulting in orbital fibroblast proliferation and release of glycosaminoglycans. The current treatments available, especially glucocorticoids, are not effective in all patients. Two cases of patients with GO treated with Sirolimus have been reported with an excellent response to the drug.

The rationale for the use of Sirolimus lies in its mechanisms of action. Sirolimus is able to inhibit T-cell activation as well as fibroblast proliferation. In addition, acts indirectly on the Insulin-Like Growth Factor-1 (IGF-1) pathway, and recent clinical trials have shown that a monoclonal antibody against the IGF-1 receptor (Teprotumumab) is effective in patients with GO. Thus, Sirolimus could be used in GO as monotherapy in patients with GO.

The aim of the present drug vs standard treatment, open-label, randomized clinical trial is to evaluate the efficacy of Sirolimus in patients with moderately severe, active GO.

54 patients (27 per group) will be randomized into two groups, A and B. Patients in group A will receive Sirolimus for 12 weeks. Patients in group B will receive methylprendnisolone for 12 weeks.

The primary objective of the study is the response of GO at 24 weeks based on a composite evaluation. The secondary Objectives will be: 1) the response of of GO at 12, 36 and 48 weeks; 2) Relapse of GO at 36 and 48 weeks (worsening compared with the 24-week evaluation); 3) The reduction of proptosis at 12, 24, 36 and 48 weeks (proportion of patients with a reduction of proptosis of at least 2 mm); 4) Reduction of the GO clinical activity score (CAS) at 12, 24, 36 and 48 weeks; 5) Quality of life (Qol) at 12, 24, 36 and 48 weeks.

The safety objectives will be adverse events, adverse drug reactions, unexpected adverse reaction, suspected unexpected adverse reactions and death, across the study and at 12, 24, 36 and 48 weeks.

DETAILED DESCRIPTION:
Study Design Phase II, randomized, adaptive, superiority, open-label, single-center, pilot clinical trial.

Fifty-four patients with moderate-to-severe and active GO will be randomized into two intervention groups, A and B, with a ratio of 1: 1. Subjects assigned to group A will receive Sirolimus for 12 weeks. Patients assigned to group B will receive a cumulative dose of 4.5 g of methylprednisolone divided into 12 weekly infusions. This treatment scheme is the clinical standard and patients would be treated with methylprednisolone in any case, even if they did not accept to participate to the study.

Enrollment duration: 24 months Study duration: 36 months Tentative start of trial: July 1st 2022

Study Population Fifty-four patients with Graves' disease and GO will be recruited during the routine clinical activity carried out at the Endocrinology Unit II of AOUP, which is a tertiary referral center for thyroid diseases.

Study Timeline

* Screening visit (2-6 weeks before the first visit)
* 1st (baseline) visit - (Time 0): randomization and administration of the first dose of trial agent
* Treatment period (week 1-week 12): daily administration of the trial agent (Sirolimus) or weekly administration of the standard treatment (methylprednisolone)
* Methylprednisolone treatment period and treatment visits (week 2-week 13); weekly methylprednisolone administrations (week 2-week 13)
* Safety visits (week 3, 5, 7, 9, 11)
* 2nd visit (week 12)
* 3rd visit (week 24)
* 4th visit (week 36)
* 5th visit (week 48)

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
2. A diagnosis of Graves' disease based on the presence of hyperthyroidism (either untreated or treated with antithyroid drugs) associated with detectable anti-thyrotropic hormone (TSH) receptor autoantibodies (TRAb). Patients must be euthyroid under control on stable medical regimen and every effort will be made to maintain the euthyroid status for the entire duration of the clinical trial
3. A moderate-to-severe GO, defined as the presence of at least one of the following criteria: an exophthalmos ≥2 mm compared with normal values for sex and race; presence of inconstant to constant diplopia; a lid retraction ≥2 mm
4. Active GO: CAS (4) ≥2 out of 7 points in the most affected eye
5. GO duration ≤18 months
6. Male and female patients of age: 18-75 years
7. Creatinine values within the reference range
8. Indexes of liver function (AST, ALT, γGT, alkaline phosphatase, total and direct bilirubin) within the normal range
9. Normal blood count, absence of diseases of hematopoiesis
10. Women of childbearing potential (WOCBP, namely not in menopause or in menopause since less than two years; in all other instances women will be considered as non-WOCBP) and men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year (as indicated in Appendix) for at least 6 and 7,5 months, respectively, after the last dose of the investigational drug (see also 2014_09_HMA_CTFG_Contraception.pdf, namely the "2014 CTFG Reccommendtions related to contraception and pregnancy testing in clinical trials")
11. Compliant patients, regular follow-up possible

Exclusion Criteria:

1. Optic neuropathy
2. Treatment with glucocorticoids, other immunosuppressive drugs or selenium for the last three months
3. Previous surgery or radiotherapy for GO
4. Radioiodine treatment for hyperthyroidism over the last 3 months, as it can affect GO
5. Contraindications to Sirolimus: hypersensitivity to the active substance or to any of the excipients; use of medications interfering with the pharmacokinetic and/or pharmacodynamic properties of rapamycin (e.g. CYP3A4 inhibitors or inducers; see "prohibited therapies")
6. Contraindications to GC: hypersensitivity to the active substance or to any of the excipients; uncontrolled hypertension, uncontrolled diabetes; history of peptic ulcer; urinary infections, glaucoma, systemic fungal infections, systemic infections unless appropriate therapy is employed, idiopathic thrombocytopenic purpura, cerebral edema associated with malaria.
7. Use of medications interfering with GC or increasing the risk of GC-related adverse events (see prohibited therapies)
8. Pregnant or lactating females as determined by positive serum or urine HCG test at baseline
9. Acute or chronic liver disease
10. Relevant malignancies
11. Current and/or previous diseases of hematopoiesis
12. Recent (≤1 year) history of alcoholism or drug abuse
13. Mental illness that prevent patients from comprehensive, written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
GO overall response | 24 weeks
  Percentage of subjects with at least two of the following compared to baseline: a) Improvement in CAS by at least 1 point ; b) Improvement in exophthalmos by at least 2 mm; c) Improvement in lid aperture by at least 2 mm; d) Improvement in eye muscle ductions ≥8 degrees; e) Improvement of visual acuity by at least 0.2/1, without worsening of any of these parameters in the contralateral eye if applicable.

SECONDARY OUTCOMES:
GO overall response | 12 weeks
  Percentage of subjects with at least two of the following compared to baseline: a) Improvement in CAS by at least 1 point ; b) Improvement in exophthalmos by at least 2 mm; c) Improvement in lid aperture by at least 2 mm; d) Improvement in eye muscle ductions ≥8 degrees; e) Improvement of visual acuity by at least 0.2/1, without worsening of any of these parameters in the contralateral eye if applicable.
GO overall response | 36 weeks
  Percentage of subjects with at least two of the following compared to baseline: a) Improvement in CAS by at least 1 point ; b) Improvement in exophthalmos by at least 2 mm; c) Improvement in lid aperture by at least 2 mm; d) Improvement in eye muscle ductions ≥8 degrees; e) Improvement of visual acuity by at least 0.2/1, without worsening of any of these parameters in the contralateral eye if applicable.
GO overall response | 48 weeks
  Percentage of subjects with at least two of the following compared to baseline: a) Improvement in CAS by at least 1 point ; b) Improvement in exophthalmos by at least 2 mm; c) Improvement in lid aperture by at least 2 mm; d) Improvement in eye muscle ductions ≥8 degrees; e) Improvement of visual acuity by at least 0.2/1, without worsening of any of these parameters in the contralateral eye if applicable.
GO relapse | 36 weeks
  Percentage of subjects with worsening of GO in comparison with the 24 week evaluation. Worsening is defined as change in two of the following in at least one eye (compared to baseline): a) Worsening in CAS by at least 1 point; b) Worsening of exophthalmos (>2 mm); c) Worsening of lid aperture (>2 mm); d) Worsening of eye ductions ≥8 degrees; d) Worsening of visual acuity by at least 0.2/1
GO relapse | 48 weeks
  Percentage of subjects with worsening of GO in comparison with the 24 week evaluation. Worsening is defined as change in two of the following in at least one eye (compared to baseline): a) Worsening in CAS by at least 1 point; b) Worsening of exophthalmos (>2 mm); c) Worsening of lid aperture (>2 mm); d) Worsening of eye ductions ≥8 degrees; d) Worsening of visual acuity by at least 0.2/1
Change in exophthalmos | 12 weeks
  Percentage of subjects with a reduction greater than or equal to 2 mm compared with the baseline evaluation in the study eye, without worsening in the contralateral eye
Change in exophthalmos | 24 weeks
  Percentage of subjects with a reduction greater than or equal to 2 mm compared with the baseline evaluation in the study eye, without worsening in the contralateral eye
Change in exophthalmos | 36 weeks
  Percentage of subjects with a reduction greater than or equal to 2 mm compared with the baseline evaluation in the study eye, without worsening in the contralateral eye
Change in exophthalmos | 48 weeks
  Percentage of subjects with a reduction greater than or equal to 2 mm compared with the baseline evaluation in the study eye, without worsening in the contralateral eye
Change in the clinical activity score (CAS) | 12 weeks
  Percentage of subjects with a reduction of CAS by at least two points in the study eye, without worsening in the contralateral eye
Change in the clinical activity score (CAS) | 24 weeks
  Percentage of subjects with a reduction of CAS by at least two points in the study eye, without worsening in the contralateral eye
Change in the clinical activity score (CAS) | 36 weeks
  Percentage of subjects with a reduction of CAS by at least two points in the study eye, without worsening in the contralateral eye
Change in the clinical activity score (CAS) | 48 weeks
  Percentage of subjects with a reduction of CAS by at least two points in the study eye, without worsening in the contralateral eye
Change in quality of life | 12 weeks
  Comparison of the quality of life scores between the two groups, determined with a questionnaire specific for GO (GO-QoL)
Change in quality of life | 24 weeks
  Comparison of the quality of life scores between the two groups, determined with a questionnaire specific for GO (GO-QoL)
Change in quality of life | 36 weeks
  Comparison of the quality of life scores between the two groups, determined with a questionnaire specific for GO (GO-QoL)
Change in quality of life | 48 weeks
  Comparison of the quality of life scores between the two groups, determined with a questionnaire specific for GO (GO-QoL)
Percentage of adverse events | 48 weeks
  Percentage of adverse events, adverse drug reactions, death across the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Cisanello-Endocrinology II, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No